CLINICAL TRIAL: NCT02290678
Title: Examining the Feasibility and Efficacy of Adventure Based Therapy as a Treatment Intevention for Depression and Anxiety.
Brief Title: Pushing Limits - Adventure: Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Margaret McKinnon, Academic Head, Mood Disorders Program, St. Joseph's Healthcare Hamilton
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Adventure_PILOT
Record Dates: First submitted 2014-11-04; First posted 2014-11-14 (Estimated); Last update posted 2015-02-20 (Estimated); Status verified 2015-02

CONDITIONS: Anxiety; Depression
Keywords: Pilot Study; Adventure-based Programming
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Participate in a two day Adventure-based Programming retreat and team building exercises.
  Interventions: Behavioral: Adventure-based Programming

INTERVENTIONS:
Behavioral: Adventure-based Programming

SUMMARY:
Team building exercises have been shown to be effective in improving an individual's ability to work within a group and build working relationships with others. Adventure Therapy assimilates team building exercises and teachings into an adventure style excursion into the wilderness or other non-typical environment. This combination of exposure and learning creates a unique experience for participants which preliminary research suggests is effective in reducing feelings of hopelessness, guilt, and shame and may increase empathy, self-concept, self-confidence, and subjects' well-being have also been shown to be improved by adventure therapy.

This study will use a series of questionnaires and interviews to determine whether an adventure based therapy is both effective and reasonable as a treatment for people with mood disorders like depression and anxiety. The objective of this study is to investigate the efficacy of adventure based therapy as a treatment intervention for outpatients with mood disorders. The investigators will observe any changes in mood, perceived self- efficacy, anxiety, self-stigma, hope, quality of life enjoyment and satisfaction, leisure motivation, and stress as a result of this intervention. As well, the investigators aim to capture participant's opinions of the program.

DETAILED DESCRIPTION:
"Adventure programming is the use of experiential and challenging approaches to education, recreation, life skills and counseling. It is the use of new, unique and relevant activities to supplement conventional learning processes. Adventure-based activities are tailored to achieve desired outcomes related to specified learning objectives. The core purpose is to intensify learning and insight by focusing on the process that occurs during challenging activities."

Adventure Based Therapy (AT) is a unique approach to traditional therapy strategies. AT is based on the philosophy of "experiential education", which is defined as "learning by doing, with reflection". The idea of experiential learning is based on the belief that learning is a result of direct experience, and learning is most effective when multiple senses are actively involved. By increasing the intensity of the mental and physical demands of learning, one can be fully engaged in the learning by simultaneously stimulating all sensory systems. Psychological research on information processing indicates that multi-sensory processing increases cognitive activity such as problem solving, processing of an experience, and memory. AT combines physical activity, social empowerment, and problem solving skills into a multi-sensory experience.

Recent literature suggests that AT can benefit patients' recovery. For example, preliminary work suggests that AT is effective in reducing feelings of hopelessness, guilt, and shame, and may increase empathy. Self-concept, self-confidence, and subjects' well-being have also been shown to be improved by AT. The concept of AT stems from the idea of team building exercises, and the notion that through participation patients experience increased group cohesion, therapeutic alliance, and communication and negotiation skills. Here, we will assess these variables in patients with mood disorders participating in AT using an extensive assessment battery. In addition, we will follow patients longitudinally to assess the durability of these effects.

The present research will be a pilot study designed to modify the protocol for the main trial. We will assess engagement in treatment by exploring participants' actual experiences and how they attribute meaning to their involvement in the therapeutic adventure based program. A qualitative research design that uses the Grounded Theory method will be used. Grounded Theory promotes a focus on individuals in real life situations and local social contexts. Qualitative interviews give participants the opportunity to have their voices or stories included in research studies as well as contribute to the development of effective treatment interventions. Feasibility of the trial will be determined by analyzing resource and economic utilization throughout the pilot.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a mood disorder and a clinician referral.

Exclusion Criteria:

-

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2015-02; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility, as measured by Number of Participants who complete the Adventure-based Programming retreat and team building exercises and Qualitative engagement feedback | Up to 2 weeks following intervention
  Interviews will be conducted with participants to determine the success in engagement of participants and the execution of the study (including allocation of staff, resources, etc.).

SECONDARY OUTCOMES:
BDI-II Score | Up to 1 week following intervention
  Difference in the score of the Beck Depression Inventory II immediately after the intervention compared to baseline immediately before intervention.
BDI-II Score | 1 month following intervention
  How well the difference in the score of the Beck Depression Inventory II is retained at 1 month compared to immediately after the intervention.
BDI-II Score | 3 months following intervention
  How well the difference in the score of the Beck Depression Inventory II is retained at 3 months compared to immediately after the intervention.
BAI Score | Up to 1 week following intervention
  Difference in the score of the Beck Anxiety Inventory immediately after the intervention compared to baseline immediately before intervention.
BAI Score | 1 month following intervention
  How well the difference in the score of the Beck Anxiety Inventory is retained at 1 month compared to immediately after the intervention.
BAI Score | 3 months following intervention
  How well the difference in the score of the Beck Anxiety Inventory is retained at 3 month compared to immediately after the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- St Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Anderson, L., Schleien, S. J., McAvoy, L., Lais, G., & Seligmann, D. (1997). Creating positive change through an integrated outdoor adventure program. Therapeutic Recreation Journal, Fourth Quarter, 214-229.
- [Background] Bandoroff, S. & Newes, S. "Coming Of Age: Evolving Field of Adventure Therapy" (2004). Association for Experiential Education. Volume 3.
- [Background] Beck, A. T., & Steer, R. A. (1990). Manual for the Beck Anxiety Inventory. San Antonio, TX: Psychological Corporation.
- [Background] BECK AT, WARD CH, MENDELSON M, MOCK J, ERBAUGH J. An inventory for measuring depression. Arch Gen Psychiatry. 1961 Jun;4:561-71. doi: 10.1001/archpsyc.1961.01710120031004. No abstract available. PMID 13688369
- [Background] Gillen, M., & Balkin, R. (2006). Adventure counseling as an adjunct to group counseling in hospital and clinical settings. Journal for Specialists in Group Work, 31(2), 153-164. doi: 10.1080/01933920500493746
- [Background] Ewert, A. W., McCormick, B. P., & Voight, A. E. (2001). Outdoor experiential therapies: Implications for TR practice. Therapeutic Recreation Journal, Second Quarter, 170-122.
- [Background] Chakravorty, D., Trunnell, E. P., & Ellis, G. D. (1995). Ropes course participation and post-activity processing on transient depressed mood of hospitalized adult psychiatric patients. Therapeutic Recreation Journal, Second Quarter, 104-113.
- [Background] Charmaz, K. (2003). Grounded Theory: Objectivist and Constructivist Methods. Strategies of Qualitative Inquiry, Denzin & Lincoln (EDS.). Sage.
- [Background] Charmaz, K. (2006). Constructing grounded theory: A practical guide through qualitative analysis, Pine Forge Press.
- [Background] Corbin, J. & Strauss, A. (2008). Basics of qualitative research: Techniques and procedures for developing grounded theory, Sage.
- [Background] Kyriakopoulos, A. (2011). How individuals with self-reported anxiety and depression experienced a combination of individual counseling along with an adventurous outdoor experience: A qualitative evaluation. Counseling and Psychotherapy Research, 11(2), 120-128. doi: 10.1080/14733145.2010.485696
- [Background] Liamputtong P. Qualitative data analysis: conceptual and practical considerations. Health Promot J Austr. 2009 Aug;20(2):133-9. doi: 10.1071/he09133. PMID 19642962
- [Background] Patton, M.Q. (2002). Qualitative Research & Evaluation Methods. (3rd edition). Thousand Oaks, CA. Sage.
- [Background] Riley, K. (2011). Effects of a collaborative outpatient therapy program on self-concept of adolescents with depression. Therapeutic Recreation Journal, 45(1), 32-46.
- See also: Directly quoted from in the project description. Gives a brief overview of Adventure Programming. — http://ct-bristol.civicplus.com/DocumentCenter/Home/View/519